CLINICAL TRIAL: NCT01047995
Title: Plasma and Intracellular Pharmacokinetics of Once Daily Darunavir/Ritonavir and Twice and Once Daily Raltegravir in HIV-infected Subjects
Brief Title: Pharmacokinetics (PK) Study of Once Daily Darunavir/Ritonavir and Twice and Once Daily Raltegravir in HIV-infected Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Dr Marta Boffito, St Stephen's AIDS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSAT 031; 2008-008321-30 (Other: EU Clinical Trials Database)
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Phase 1, all subjects (n = 24): Raltegravir 400 mg twice daily for 21 days
  Phase 2 Group 1 (n = 12): Darunavir/ritonavir 800/100 mg once daily plus raltegravir 400 mg twice daily for 14 days
  Phase 3, all subjects (n = 24): Darunavir/ritonavir 800/100 mg once daily for 14 days.
  Interventions: Drug: Raltegravir plus Darunavir/ritonavir
- Group 2 (Active Comparator): Phase 1, all subjects (n = 24): Raltegravir 400 mg twice daily for 21 days
  Phase 2,
  Group 2 (n = 12): Darunavir/ritonavir 800/100 mg once daily plus raltegravir 800 mg once daily for 14 days
  Phase 3, all subjects (n = 24): Darunavir/ritonavir 800/100 mg once daily for 14 days.
  Interventions: Drug: Raltegravir plus Darunavir/ritonavir

INTERVENTIONS:
Drug: Raltegravir plus Darunavir/ritonavir — Phase 1, all subjects (n = 24): Raltegravir 400 mg twice daily for 21 days
  Phase 2 Group 1 (n = 12): Darunavir/ritonavir 800/100 mg once daily plus raltegravir 400 mg twice daily for 14 days
  Phase 3, all subjects (n = 24): Darunavir/ritonavir 800/100 mg once daily for 14 days.
  Other Names: darunavir = TMC114; ritonavir = Norvir trade name; raltegravir = MK-0518, brand name Isentress
  Arms: Group 1
Drug: Raltegravir plus Darunavir/ritonavir — Phase 1, all subjects (n = 24): Raltegravir 400 mg twice daily for 21 days
  Phase 2
  Group 2 (n = 12): Darunavir/ritonavir 800/100 mg once daily plus raltegravir 800 mg once daily for 14 days
  Phase 3, all subjects (n = 24): Darunavir/ritonavir 800/100 mg once daily for 14 days.
  Other Names: darunavir = TMC114; ritonavir = Norvir trade name; raltegravir = MK-0518, brand name Isentress
  Arms: Group 2

SUMMARY:
The study aims to help us understand if the HIV drugs darunavir (taken with ritonavir) and raltegravir will affect each other when they are given at the same time.

The purpose of the study is to assess the pharmacokinetics (how a drug is absorbed, distributed and eliminated from your body) of darunavir and ritonavir when these are taken with and without raltegravir.

The duration of the study will be up to 50 days plus a screening visit which will take place up to 4 weeks prior to the start of the study, and a follow up visit which takes place 1-2 weeks after the last dose of study medication.

Subjects will continue to take 2 of their usual drugs (those called nucleoside reverse transcriptase inhibitors -NRTI) throughout the study.

For the first 21 days subjects will take their usual NRTI plus raltegravir 400mg twice daily. After this, subjects will also receive either:

Group 1) Darunavir/ritonavir 800mg/100mg once daily AND raltegravir 400mg twice daily or Group 2) Darunavir/ritonavir 800mg/100mg once daily AND raltegravir 800mg once daily

Subjects will take this regimen for 14 days. Subjects will be randomly allocated to either Group 1 or 2. You will have an equal (50/50) chance of being allocated to Group 1 or 2.

DETAILED DESCRIPTION:
The integrase inhibitor raltegravir has shown to a potent new agent for the treatment of HIV infection.

When raltegravir and darunavir/ritonavir have been combined in the Benchmark studies, they provided an excellent virological response in highly experienced patients.

Darunavir once daily use is increasing due to patients' preference for once daily regimens.

Raltegravir has not shown any pharmacokinetic/pharmacodynamic relationship and doses of 100 to 400 mg twice daily have shown similar virological responses. This may be due to intracellular drug accumulation.

However, data on the use of darunavir/r plus raltegravir once daily and on raltegravir intracellular concentrations are not available.

Whether raltegravir is efficacious when administered once daily is unknown. However, concentrations higher the IC95 of 33nM have been associated to a favourable virological response.

Therefore, we would like to investigate the plasma and intracellular pharmacokinetics of darunavir/ritonavir and raltegravir when co-administered once daily in order to provide further data to support the use of these agents once daily, patients' preferred dosing schedule.

Pharmacogenetics holds promise in HIV treatment because of the complexity and potential toxicity of multi antiretroviral drug therapies that are prescribed for long periods. Thus far, few candidate genes have been examined for a limited number of allelic variants, but a number of confirmed associations have already emerged.

From a public health perspective, as antiretroviral medications become increasingly available to racially and ethnically diverse populations worldwide, understanding the genetic structures of each population may allow us to anticipate the impact of adverse responses, even in groups that were not represented in drug registration trials.

The existing literature on pharmacogenetic determinants of antiretroviral drug exposure, drug toxicity, as well as genetic markers associated with the rate of disease progression underline the recent advances which occurred in the past few years.

However, it is expected that larger-scale comprehensive genome approaches will profoundly change the landscape of knowledge in the future. Additional studies are needed to assess the implications for long-term responses to antiretroviral agents.

For this reason we plan to collect a single blood sample from each participant in our intensive pharmacokinetic studies, such as this one, in order to be able to investigate the association between genetic polymorphisms in drug disposition genes (such as those encoding for cytochrome P450 isoenzymes or transmembrane transporters) and drug exposure. A candidate gene approach will be utilised to examine loci of interest. This procedure will provide potentially important information on genetic influences on plasma drug concentrations and give insight into how to improve the management of HIV-infected patients by individualising therapy. These studies will not be powered for genetic associations but will enable us to build a data base of genotype-phenotype. Prospective genetic studies would need to be planned based on these preliminary data.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria within 28 days prior to the baseline visit:

1. The ability to understand and sign a written informed consent form, prior to participation in any screening procedure and must be willing to comply with all study requirements.
2. Male or non-pregnant, non-lactating females.
3. Between 18 to 65 years, inclusive.
4. Documented HIV-1 infection and plasma HIV RNA at screening visit below 400 copies/mL.

   (Note retesting of screening viral load is allowed).
5. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study.
6. CD4 count > 100 at screening (Note retesting of screening CD4 count is allowed).
7. Receiving an antiretroviral regimen including two NRTIs and an NNRTI or a boosted protease inhibitor or an integrase inhibitor, without any history of virological failure (history of drug switches is allowed only if the reason was tolerability/toxicity/convenience of dosing).
8. Agrees not to change regimen, outside the study recommendations, from baseline until end of the treatment period unless this is medically indicated as decided by the treating physician.

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria are not to be enrolled in this study.

1. Any serious or active medical or psychiatric illness which, in the opinion of the investigator, would interfere with subject treatment, assessment, or compliance with the protocol. This would include any active clinically significant renal, cardiac, hepatic, pulmonary, vascular, metabolic disorders or malignancy.
2. Have a body mass index (BMI) >35
3. Presence of any current active AIDS defining illness (Category C conditions according to the CDC Classification System for HIV Infection 1993) with the following exceptions:

   • Stable cutaneous Kaposi's Sarcoma
4. Clinically relevant alcohol or drug use (positive urine drug screen, with the exception of cannabinoids) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study.
5. The use of disallowed concomitant therapy (See Concomitant Medication and treatment, section 5.2).
6. Females of childbearing potential without the use of effective non-hormonal birth control methods or not willing to continue practicing these birth control methods for at least 14 days after the end of the treatment period.
7. Previous allergy to any of the constituents of the pharmaceuticals administered in this trial.
8. Subjects with clinical or laboratory evidence of significantly decreased hepatic or renal function (as determined by the principal investigator).
9. Exposure to any investigational drug or placebo within 4 weeks of first dose of study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Steady state plasma and intracellular concentrations of darunavir/ritonavir once daily with and without raltegravir and raltegravir twice and once daily | 50 days

SECONDARY OUTCOMES:
Safety and tolerability of darunavir/ritonavir and raltegravir when co-administered to HIV-infected subjects | 50 days
Association between genetic polymorphisms in drug disposition genes and drug exposure | 50 days

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Dr, Principal Investigator — St Stephen's AIDS Trust
Locations (2):
- United Kingdom (2):
  - St Stephen's Centre, Chelsea and Westminster Hospital NHS Foundation Trust, London, London
  - St Stephens Centre, Chelsea & Westminster Hospital, London